CLINICAL TRIAL: NCT02342847
Title: Observational Cohort Study of Health-related Quality of Life in Patients Initiating Treatment With Chemotherapy for Metastatic Pancreatic Cancer
Brief Title: Observational Study of Quality of Live in Patients With Metastatic Pancreatic Cancer
Acronym: aLIVE
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-CPM-2014-01
Record Dates: First submitted 2014-12-30; First posted 2015-01-21 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pateints with metastatic pancreatic cancer: Patients diagnosed with metastatic pancreatic cancer confirmed histologically or cytologically, who will be treated with chemotherapy as first-line treatment of metastatic pancreatic cancer.
  This study is designed to observe patients treated in routine clinical practice, without the exclusion limitations of a clinical trial. The decision to treat patients will be performed prior to the decision to include the patient in the study.
  The follow-up of patients will be performed according to standard clinical practice of each site
  Interventions: Other: N/A (non-interventional study)

INTERVENTIONS:
Other: N/A (non-interventional study)

SUMMARY:
This is an observational, post-authorization, prospective follow-up, multi-centre, national study designed to describe the spectrum of health-related quality of life in patients with metastatic pancreatic cancer previously untreated with chemotherapy This study is designed to observe patients treated in routine clinical practice, without the exclusion limitations of a clinical trial. Patients will be enrolled in 7 Spanish sites. In all cases, the decision to treat patients will be performed prior to the decision to include the patient in the study.

Given the observational nature of the study, follow-up of patients will be performed according to standard clinical practice of each site.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Patients diagnosed with metastatic pancreatic cancer confirmed histologically or cytologically
* Patients with Karnofsky index ≥ 70 previously untreated with chemotherapy.
* Patients with life expectancy ≥ 6 months.
* Patients who will be treated with chemotherapy as first-line treatment for metastatic pancreatic cancer.*
* Informed consent in writing or orally before witnesses.

  * The decision to prescribe any treatment will be clearly dissociated from the patient's inclusion in the study. Therefore, the choice of therapeutic strategy will be made according to usual clinical practice and independently by the doctor before assessing the possible involvement of the patients in the study and their corresponding inclusion in it

Exclusion Criteria:

* Pregnant or breastfeeding.
* Patients who are participating in an interventional clinical trial.
* Patients who refuse to participate in this study.
* Patients who have no ability to understand and respond to questions related to their health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be treated with any of the first line chemotherapy treatments at the participating site approved for the treatment of Metastasic Pancreatic Cancer (MPC) will be included consecutively according to the criteria set.
  Therefore, the choice of therapeutic strategy will be made according to usual clinical practice and independently by the doctor before assessing the possible involvement of the patients in the study and their corresponding inclusion in it.
  The patients selected for the study must meet all inclusion criteria and none of the exclusion.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Patients with mild improvement in Quality of life questionnaire - Current standard version 3.0 (EORTC QLQ-C30) scoring | Up to 18 months
  Number of participants with mild improvement. Mild improvement in QoL : (increased from ≥ 5 to <10 points), moderate (increase of between ≥ 10 and <20 points), and high (increase ≥ 20 points) in EORTC QLQ-C30) scoring.
Patients with mild impairment of EORTC QLQ-C30 scoring | Up to 18 months
  Number of participants with mild impairment. Mild impairment of QoL (decrease from ≥ 5 to <10 points), moderate (decrease from ≥ 10 and <20 points), and severe (decrease ≥ 20 points) in EORTC QLQ-C30 scoring); mean time to improvement of Quality of Life (QoL) of mild, moderate and high in EORTC QLQ-C30 scoring
Patients with moderate improvement in EORTC QLQ-C30 scoring | Up to 18 months
  Number of participants with moderate improvement. Mild improvement in QoL (increased from ≥ 5 to <10 points), moderate (increase of between ≥ 10 and <20 points), and high (increase ≥ 20 points) in EORTC QLQ-C30) scoring.
Patients with moderate impairment of EORTC QLQ-C30 scoring | Up to 18 months
  Number of participants with moderate impairment.Mild impairment of QoL (decrease from ≥ 5 to <10 points), moderate (decrease from ≥ 10 and <20 points), and severe (decrease ≥ 20 points) in EORTC QLQ-C30 scoring); mean time to improvement of QoLof mild, moderate and high in EORTC QLQ-C30 scoring
Patients with high improvement in EORTC QLQ-C3 scoring | Up to 18 months
  Number of participants with high improvement. Mild improvement in QoL (increased from ≥ 5 to <10 points), moderate (increase of between ≥ 10 and <20 points), and high (increase ≥ 20 points) in EORTC QLQ-C30) scoring.
Patients with high impairment of EORTC QLQ-C30 scoring | Up to 18 months
  Number of participants with high impairment. Mild impairment of QoL (decrease from ≥ 5 to <10 points), moderate (decrease from ≥ 10 and <20 points), and severe (decrease ≥ 20 points) in EORTC QLQ-C30 scoring); mean time to improvement of QoLof mild, moderate and high in EORTC QLQ-C30 scoring
Impairment of mild EORTC QLQ-C30 score | Up to 18 months
  Time from enrolment to the first observation of a definite impairment of mild EORTC QLQ-C30 score (decrease from ≥ 5 to <10 points without further improvement ≥ 5 points)
Deterioration of Moderate EORTC QLQ-C30 Score | Up to 18 months
  The time from enrollment to the first observation of a definite deterioration of moderate EORTC QLQ-C30 score (decrease from ≥ 10 and <20 points without further improvement ≥ 10 points)
Deterioration of severe EORTC QLQ-C30 | Up to 18 months
  Time from enrolment to the first observation of a definite deterioration of moderate EORTC QLQ-C30 score (decrease from ≥ 10 and <20 points without further improvement ≥ 10 points)
Definite deterioration of moderate EORTC QLQ-C30 Score | Up to 18 months
  Percentage of Time from enrollment to the first observation of a definite deterioration of moderate EORTC QLQ-C30 score (decrease from ≥ 10 and <20 points without further improvement ≥ 10 points)
Mild/moderate/severe decline in EORTC QLQ-C30 | Up to 18 months
  Number of patients with mild/moderate/severe decline in EORTC QLQ-C30 on the 30th day, 2nd month, 3rd month, 4th month, 5th month and 6th month.
Patients with mild/moderate/high improvement in EORTC QLQ-C30 | Up to 18 months
  Percentage of patients with mild/moderate/high improvement in EORTC QLQ-C30 on the 30th day, 2nd month, 3rd month, 4th month, 5th month and 6th month.
Deterioration of severe QLQ-C30 | Up to 18 months
  Time from enrolment to the first observation of a definite deterioration of moderate EORTC QLQ-C30 score (decrease from ≥ 10 and <20 points without further improvement ≥ 10 points)
Change from baseline of the EuroQoL Five Dimensions Questionnaire (EQ-5D). | Up to 6 months
  Change from baseline of the EQ-5D questionnaire at 15 days, 4 weeks, 2 months, 3rd month, 4th month, 5th month and 6th month
Change from baseline of the Karnofsky index | Up to 6 months
  Change from baseline of Karnofsky index at 15 days, 4 weeks, 2 months, 3rd month, 4th month, 5th month and 6th month.

SECONDARY OUTCOMES:
Feasibility of using the EORTC QLQ-C30 and EQ-5D questionnaires | Up to 6 months
  Number of missing EORTC QLQ-C30 and EQ-5D questionnaires at 15 days, 4 weeks, 2 months, 3rd month, 4th month, 5th month and 6th month.
Average variation of Karnofsky index versus EORTC QLQ-C30 score | Up to 6 months
  Average variation of Karnofsky index regarding patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score.
Percentage of improved Karnofsky index | Up to 18 months
  Percentage of patients with improved Karnofsky basal index per month of treatment
Average variation of Karnofsky index versus EQ-5D score | Up to 6 months
  Average variation of Karnofsky index regarding patients with impairment or improvement of EQ-5D score.(0.1, 0.2, 0.3, 0.4 and 0.5 variation)
Percentage of improved Karnofsky index | Up to 6 months
  Percentage of patients with improved Karnofsky basal index per month of treatment
Percentage of worse Karnofsky index | Up to 6 months
  Percentage of patients with worse Karnofsky basal index per month of treatment
Mean of improvement of Karnofsky index | Up to 6 months
  Mean time to improvement of Karnofsky index from baseline
Mean of deterioration of Karnofsky index | Up to 6 months
  Mean time to deterioration of Karnofsky index in patients who have previously improved after treatment.
Weight variation | Up to 6 months
  Change in weight during treatment observation period (maximum 6 months). This outcome wil be measured overall and per group of patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score
Number of patients who use Painkillers during treatment observation period (maximum 6 months) | Up to 6 months
  Number of patients who use Painkillers during treatment observation period (maximum 6 months) with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score.
Number of patients who use analgesics during treatment observation period (maximum 6 months). | Up to 6 months
  Number of patients who use analgesics during treatment observation period (maximum 6 months) with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score.
Duration of treatment | Up to 18 months
  Average duration of treatment with chemotherapy for metastatic pancreatic cancer.
Average dose of treatment (minimum, maximum) | Up to 18 months
  Average dose (minimum, maximum) of the treatment with chemotherapy for metastatic pancreatic cancer.
Delayed/Reduced dose treatment | Up to 18 months
  Number of patients with delayed dose or with reduced dose . This outcome wil be measured overall and per group of patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score
Rate response based on the treatment given. | Up to 18 months
  Rate response (RR) wil be measured overall and per group of patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score
Response to treatment determined by (Response Evaluation Criteria in Solid Tumors )RECIST v.1.1. | Up to 18 months
  Response to treatment (RT) of the disease determined by RECIST v.1.1. . based on the treatment given This outcome wil be measured overall and per group of patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score
Overall survival determined by RECIST v.1.1. | Up to 30 months
  Overall survival (OS) of the disease determined by RECIST v.1.1. This outcome wil be measured overall and per group of patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score
Progression-free survival determined by RECIST v.1.1 | Up to 30 months
  Progression-free survival (PFS) of the disease determined by RECIST v.1.1. based on the treatment given. This outcome wil be measured overall and per group of patients with mild, moderate and high impairment and mild, moderate and severe improvement of EORTC QLQ-C30 score
Hematologic toxicity | Up to 30 months
  Number of participants with Grade 3-4 hematologic toxicity
Radiological examinations | Up to 18 months
  Number of radiological examinations per patient during treatment.
Laboratory assessments | Up to 18 months
  Number of laboratory assessments per patient during treatment
Physical examinations | Up to 18 months
  Number of physical examinations per patient during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Pellín, MD, Study Director — Celgene Spain
Locations (12):
- Spain (12):
  - Hospital Universitario Burgos, Burgos, Castille and León
  - Complejo Asistencial León, León, Castille and León
  - Hospital del Bierzo, León, Castille and León
  - Hospital Universitario Salamanca, Salamanca, Castille and León
  - Germans Trias i Pujol, Badalona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Vall d´Hebron, Barcelona, Catalonia
  - Hospital Universitario Josep Trueta de Girona, Girona, Catalonia
  - Hospital Duran I Reynals (ICO Bellvitge), L'Hospitalet de Llobregat, Catalonia
  - Hospital San Joan Reus, Reus, Catalonia
  - Hospital de Sabadell ( Parc Taulí), Sabadell, Catalonia
  - Hospital Santa Creu i Sant Pau, Barcelona